CLINICAL TRIAL: NCT04833829
Title: Cross-disciplinary HIV Integrated Mental Health Support (CHIMES) Intervention
Brief Title: Cross-disciplinary HIV Integrated Mental Health Support Intervention
Acronym: CHIMES
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Sophia Hussen, Associate Professor, Emory University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00000560; R34MH124638 (NIH)
Record Dates: First submitted 2021-04-04; First posted 2021-04-06 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Human Immunodeficiency Virus; HIV Infections
Keywords: Mental health
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections; Psychological Well-Being | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Clinic Patients During the Pre-implementation Period (Active Comparator): Patients visiting one of the study clinics prior to implementation of the CHIMES intervention. The Baseline time period consists of study Months 1 - 12. Data are retroactively abstracted from medical records of patients who had clinic visits that occurred between January 1, 2019 and December 31, 2019.
  Interventions: Behavioral: Standard of Care
- Clinic Patients During the Implementation Period (Experimental): Patients visiting one of the study clinics during the Implementation period of the CHIMES intervention. Data will be abstracted from medical records of visits that occur during study Months 13 - 27.
  Interventions: Behavioral: CHIMES Intervention
- Clinic Patients During the Maintenance Period (Experimental): Patients visiting one of the study clinics during the Maintenance period of the CHIMES intervention. Data will be abstracted from medical records of visits that occur during study Months 28 - 33.
  Interventions: Behavioral: CHIMES Intervention

INTERVENTIONS:
Behavioral: CHIMES Intervention — There are six components to the intervention:
  1. Posters and other print materials to prompt providers and patients to discuss MH care engagement.
  2. Brief verbal scripts to help HIV providers facilitate patient MH engagement and discuss barriers to MH utilization.
  3. Expanded MH screening procedures, including at initial intake.
  4. Case management, emphasizing MH care engagement.
  5. Interactive trainings for all HIV providers on MH needs, screening/treatment, and barriers to MH service utilization specific to YB-GBMSM.
  6. Regular case review meetings.
  Arms: Clinic Patients During the Implementation Period; Clinic Patients During the Maintenance Period
Behavioral: Standard of Care — The standard of care practices of referring patients to mental health services of the clinic during Months 1 - 12 of the study.
  Arms: Clinic Patients During the Pre-implementation Period

SUMMARY:
The proposed project seeks to develop and test an intervention to improve engagement in HIV and mental health care for young Black gay, bisexual and other men who have sex with men (YB-GBMSM) in Ryan White clinics.

DETAILED DESCRIPTION:
Young Black gay, bisexual and other men who have sex with men (YB-GBMSM) are disproportionately impacted by HIV, with suboptimal rates of engagement across the HIV Continuum of Care (HIV-CoC). Mental health (MH) comorbidities contribute to poor HIV care engagement for many YB-GBMSM; however, effective treatment for these conditions is hindered by barriers including logistical challenges, medical mistrust, and MH stigma.

The Ryan White Care act supports integration of HIV and MH services; however, preliminary studies demonstrate low rates of MH referrals and MH care engagement among YB-GBMSM living with HIV, even in these ostensibly integrated care settings. The objective of this study is to develop and implement CHIMES (Cross-disciplinary HIV Integrated with Mental Health Support), a clinic- and provider-level intervention to improve HIV-MH care integration and MH care engagement among YB-GBMSM attending Ryan White clinics.

The rationale for this study is that efforts to improve integration of services, particularly if they are culturally tailored, are likely to increase MH and HIV care engagement for YB-GBMSM. The proposed study will pursue two specific aims: (1) to develop the CHIMES intervention; and (2) to conduct a hybrid type 2 implementation-effectiveness pilot trial of CHIMES in two Health Resources and Services Administration (HRSA)/Ryan White-funded clinics in Atlanta, Georgia - a city in the heart of the Southern HIV epidemic.

For the first aim, the researchers will work collaboratively with provider and patient stakeholders, adapt existing evidence-based interventions, and build on formative data to refine intervention content, informed by the Capability- Opportunity-Motivation-Behavior (COM-B) Model. For the second aim, the researchers will implement CHIMES in the two clinic settings and conduct a mixed-methods assessment in which continuous data collection informed by the Reach, Effectiveness, Adoption, Implementation, Maintenance (RE-AIM) framework will be used to evaluate effectiveness and implementation processes.

The effectiveness of the CHIMES intervention will be measured by change in HIV and MH care engagement before, during, and after CHIMES implementation. The researchers will abstract clinic-level aggregate data to characterize change in HIV-CoC and MH care engagement outcomes for YB-GBMSM.

ELIGIBILITY:
Inclusion Criteria:

* young Black gay, bisexual and other men who have sex with men (YB-GBMSM) living with HIV
* patient at Grady Health System Infectious Disease Program or Emory University Hospital Midtown Infectious Disease Clinic

Exclusion Criteria:

* none

Ages: 18 Years to 29 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 850 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Number of Mental Health Visits | Baseline (Months 1-12) up to Month 33
  The number of mental health visits by clinic patients during each study time period.
Percentage of Mental Health Visits by YB-GBMSM | Baseline (Months 1-12) up to Month 33
  The percentage of mental health visits by YB-GBMSM clinic patients during each study time period.
Number of Patients Attending Two HIV Care Visits | Baseline (Months 1-12) up to Month 33
  The number of patients who come to two HIV Care visits in a 12 month period, during each study time period.
Number of Patients with HIV RNA Viral Suppression | Baseline (Months 1-12) up to Month 33
  The number of patients with HIV RNA less than 200 Copies, during each study time period.
Number of Mental Health Care Referrals | Baseline (Months 1-12) up to Month 33
  The number of referrals to mental health care during a 12 month period, during each study time period.
Percentage of Mental Health Referrals for YB-GBMSM | Baseline (Months 1-12) up to Month 33
  The percentage of mental health referrals by YB-GBMSM clinic patients during each study time period.

CONTACTS AND LOCATIONS:
Overall Officials: Sophia Hussen, MD, MPH, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Grady Infectious Diseases Clinic (Ponce Clinic), Atlanta, Georgia
  - Emory Midtown Hospital Infectious Disease Outpatient Clinic, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data will be made available to other researchers, using established public repositories.
Supporting Information: Study Protocol, SAP
Time Frame: Participant data will be made available for sharing after publication of this study.
Access Criteria: Data will be available to other researchers using established public repositories.

DOCUMENTS (1):
  • Informed Consent Form (2020-06-01): https://cdn.clinicaltrials.gov/large-docs/29/NCT04833829/ICF_000.pdf